CLINICAL TRIAL: NCT05682352
Title: A Randomized, Double-Blind, Placebo-Controlled, Single- And Multiple Ascending Dose Trial To Evaluate The Safety, Tolerability, And Pharmacokinetics Of Leo 158968 In Healthy Subjects
Brief Title: Investigating the Safety of LEO 158968 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: LP0189-2242; 2022-002768-65 (EudraCT Number); U1111-1285-9850 (Other: WHO (World Health Organization))
Record Dates: First submitted 2023-01-04; First posted 2023-01-12 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; LEO 158968

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LEO 158968 Single Ascending Dose (SAD) Cohorts (Experimental): Participants will receive a single dose of LEO 158968 or matching placebo via an intravenous (IV) infusion or subcutaneous (SC) injection. The dose of LEO 158968 will be increased per cohort.
  Interventions: Drug: LEO 158968; Drug: Placebo
- LEO 158968 Multiple Ascending Dose (MAD) Cohorts (Experimental): Participants will receive 5 once weekly (QW) doses of LEO 158968 or matching placebo via a SC injection.
  Interventions: Drug: LEO 158968; Drug: Placebo

INTERVENTIONS:
Drug: LEO 158968 — IV infusion or SC injection
  Arms: LEO 158968 Single Ascending Dose (SAD) Cohorts
Drug: Placebo — IV infusion or SC injection
  Arms: LEO 158968 Single Ascending Dose (SAD) Cohorts
Drug: LEO 158968 — SC injection
  Arms: LEO 158968 Multiple Ascending Dose (MAD) Cohorts
Drug: Placebo — SC injection
  Arms: LEO 158968 Multiple Ascending Dose (MAD) Cohorts

SUMMARY:
The purpose of this study is to investigate what side effects the new compound LEO 158968 might cause and how well it is tolerated when it is used by healthy participants. It will also investigate how quickly and to what extent LEO 158968 is distributed and eliminated from the body and if LEO 158968 causes the body to make antibodies.

In the single ascending dose (SAD) cohorts, participants will receive escalating doses of LEO 158968 if the safety and tolerability results of the initial participants up to 48 hours (or 4 days for SC dosing) following dosing are acceptable to the Investigator.

In the multiple ascending dose (MAD) cohorts, the dose of LEO 158968 will be determined based on results derived from the earlier SAD cohorts and additional preclinical data from a 5-week good laboratory practice (GLP) cynomolgus monkey toxicology study.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 60 years, inclusive, at screening
2. Sex: Male or female
3. Body mass index: 18.0 kg/m^2 to 32.0 kg/m^2, inclusive, at screening
4. Health status: In good health as judged by the Investigator based on medical history, physical examination, electrocardiogram (ECG), hematology, biochemistry, and urinalysis.

Exclusion Criteria:

A participant who meets any of the following exclusion criteria will not be eligible for inclusion in the study:

1. Male participants sexually active with a woman of childbearing potential who are not willing to use a barrier method of contraception (eg, condom) from the time of first dose of investigational medicinal product (IMP) until 16 weeks after the last dose, in conjunction with this female partner using a highly effective form of contraception.
2. Female participants who are pregnant, lactating, or planning to become pregnant during the time of the trial.
3. Participants with any surgical or medical condition which might significantly alter the distribution, metabolism, or excretion of any drug.
4. Positive polymerase chain reaction (PCR) test for coronavirus disease-19 (COVID-19) on Day -1, or contact with COVID-19 positive (or suspected) persons within 14 days prior to first dose.
5. ECG with QT-interval corrected for heart rate (QTc) using Fridericia's formula (QTcF) >450 msec for men, >460 msec for women, confirmed by repeat measurement at screening.
6. Treatment with any prescribed or nonprescribed systemic or topical medication within 7 days prior to the first dose of IMP (excluding paracetamol; including herbal remedies), unless, in the opinion of the Investigator and the Sponsor, the medication will not interfere with the trial procedures or compromise safety.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Number of Treatment-emergent Adverse Events (TEAEs) Reported for Each Participant | Day 1 to Day 113
  Any clinically significant changes from baseline in clinical laboratory parameters, vital signs including systolic and diastolic blood pressure, and abnormal clinically significant findings from physical examinations following first dose will be recorded as TEAEs.

SECONDARY OUTCOMES:
Area Under the Serum Concentration-time Curve from Time 0 to Infinity (AUC0-∞) of LEO 158968 | Day 1 to Day 85
Area Under the Serum Concentration-time Curve from 0 Hours to 168 Hours (AUC0-168h) of LEO 158968 | Day 1 to Day 85
Area Under the Serum Concentration-time Curve from t=0 to t (AUC0-t) of LEO 158968 | Day 1 to Day 85
  Where t corresponds to the last observed quantifiable concentration calculated by the linear up - logarithmic down trapezoidal rule.
Serum Concentration Observed at 168 Hours Post-dose (C168h) of LEO 158968 | Day 1 to Day 85
Maximum Observed Serum Concentration (Cmax) of LEO 158968 | Day 1 to Day 85
Apparent Terminal Half-life (t1/2) of LEO 158968 | Day 1 to Day 85
Time of Last Quantifiable Concentration (tlast) of LEO 158968 | Day 1 to Day 85
Time of Cmax (tmax) of LEO 158968 | Day 1 to Day 85
Area Under the Serum Concentration-time Curve Over the Dosing Interval τ (ie, 168 hours) (AUCτ) of LEO 158968 | Day 1 to Day 113
AUC0-t of LEO 158968 | Day 1 to Day 113
Trough Serum Concentration Observed at the End of a Dosing Interval (168 hours post-dose) (Cτ) of LEO 158968 | Day 1 to Day 113
Cmax of LEO 158968 | Day 1 to Day 113
t1/2 of LEO 158968 | Day 1 to Day 113
tlast of LEO 158968 | Day 1 to Day 113
tmax of LEO 158968 | Day 1 to Day 113
Number of Participants with Antidrug Antibodies (ADA) | Day 1 to Day 113

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (1):
- LEO Pharma Investigational Site, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No